CLINICAL TRIAL: NCT07199569
Title: A Randomized, Double-blind, Phase 2b Comparability Trial in Adults 18 to 49 Years of Age to Assess Immunogenicity, Safety, and Reactogenicity of the MVA-BN Vaccine Manufactured in Different Production Cells
Brief Title: Comparability Trial of the MVA-BN Vaccine Manufactured in Different Production Cells
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: POX-MVA-046
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Monkeypox (Mpox)
MeSH Terms: conditions — Mpox, Monkeypox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): MVA-BN (CEF)
  Interventions: Biological: Jynneos
- Group 2 (Experimental): MVA-BN (Quail)
  Interventions: Biological: MVA-BN (Quail)

INTERVENTIONS:
Biological: Jynneos — MVA-BN manufactured in primary CEF cells. MVA-BN (CEF) vaccine contains 0.5 × 10E8 to 3.95 × 10E8 Inf.U and is an LF suspension to be administered subcutaneously into the deltoid muscle of the upper arm (preferably the nondominant arm). Participant will receive 2 doses 4 weeks apart (Day 1 and Day 29).
  Arms: Group 1
Biological: MVA-BN (Quail) — MVA-BN manufactured in CCX.E10 quail cell line. Vaccine contains 0.5 × 10E8 to 3.95 × 10E8 Inf.U. and is a LF suspension to be administered subcutaneously into the deltoid muscle of the upper arm (preferably the nondominant arm). Participant will receive 2 doses 4 weeks apart (Day 1 and Day 29).
  Arms: Group 2

SUMMARY:
andomized, double-blind, phase 2b trial to assess comparability in immunogenicity, safety, and reactogenicity of MVA-BN vaccine manufactured in primary chicken

embryo fibroblast (CEF) cells and the CCX.E10 quail cell line in adults

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 49 years of age
2. Informed consent form (ICF) signed and dated by the participant after reading the form and being advised of the risks and benefits of the trial in a language understood by the participant and before performance of any trial-specific procedures
3. General good health, without clinically relevant medical illness, physical exam findings, or laboratory abnormalities, as determined by the investigator that would interfere with the trial
4. Body mass index (BMI) ≥18.5 and ≤35 (calculated as [body weight in kg]/[body height in m]2 )
5. Agreement by female participants of childbearing potential and male participants who are sexually active with a female partner of childbearing potential to use a highly effective method of birth control from at least 30 days prior to administration of the MVA-BN vaccine until 30 days after last vaccination

   1. Medically acceptable methods of contraception that may be used by the participant and/or partner include combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), combined use of 2 barrier birth control methods (male condom with female diaphragm, male condom with cervical cap), bilateral tubal occlusion, vasectomy, or abstinence (acceptable only if refraining from heterosexual intercourse during the entire period of 30 days prior to administration of the MVA-BN vaccine until 30 days after last vaccination
   2. Female participants or partners are not considered to be of childbearing potential if they are at least 1 year postmenopausal

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Acute or chronic condition that, in the opinion of the investigator, would render the trial procedures unsafe or would interfere with the evaluation of responses including, but not limited to, neurologic, cardiovascular, respiratory, hepatic, hematologic, rheumatologic, endocrine, gastrointestinal, renal, autoimmune, or immunosuppressive conditions
3. History of or active autoimmune disease (vitiligo or thyroid disease requiring thyroid replacement are not exclusions), history of Guillain-Barré syndrome or Reye's syndrome
4. Known immunodeficiency syndrome or known or suspected impairment of immunologic functions including, but not limited to, clinically significant liver disease, diabetes mellitus type I, or moderate to severe kidney impairment; HIV infection under stable HAART regimen (no change within the last 3 months) and CD4 count is >500/µL is not considered immunodeficient
5. Known or reported previous smallpox vaccination or vaccination with any licensed or investigational poxvirus-based vaccine
6. History of monkeypox, cowpox, or vaccinia infection
7. Close contact in the 3 weeks prior to signing the ICF with anyone known to have mpox
8. History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision at least 6 months prior to screening that is considered to have achieved cure
9. Clinically significant mental disorder not adequately controlled by medical treatment
10. Active or recent (within 6 months before screening) chronic alcohol abuse and/or intravenous and/or nasal drug abuse
11. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, eg, tris(hydroxymethyl)-amino methane, including history of allergic asthma
12. Known allergy to aminoglycosides or quinolones
13. History of anaphylaxis or severe allergic reaction to any vaccine
14. Receipt of or plans to receive any licensed live vaccine from 30 days prior to the trial vaccination until 30 days after last trial vaccination
15. Receipt of or plans to receive any licensed nonlive vaccine from 14 days prior to the trial vaccination until 14 days after last trial vaccination
16. Use of any investigational or nonregistered agent within 30 days prior to vaccination or plans to receive an investigational agent during the trial
17. Recent blood donation (including platelets, plasma, and red blood cells) within 4 weeks prior to screening, or planned blood donations during the active trial period
18. Chronic systemic administration (defined as more than 14 days) of >5 mg prednisone (or equivalent)/day or any other immune-modifying drugs from 3 months prior to the first trial vaccination to the visit at the end of the active trial period (use of topical, inhaled, ophthalmic, and nasal glucocorticoids is allowed)
19. History of organ transplantation whether or not chronic immunosuppressive therapy is being administered
20. Abnormal troponin I level >upper limit of normal (ULN)
21. Administration or planned administration of immunoglobulins and/or any blood products from 3 months prior to the first trial vaccination until the visit at the end of the active trial period (packed red blood cells given for an emergency indication in an otherwise healthy person and not required as ongoing treatment is not exclusionary [eg, packed red blood cells given in an emergency during elective surgery])
22. History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, significant arrhythmia with or without corrective/ablative surgery, or any other heart condition under the care of a doctor
23. Employment with the investigator or trial site, with direct involvement in the proposed trial or other studies under the direction of that investigator or trial site, or relationship to the investigator or trial site employee
24. Relationship with Bavarian Nordic as an employee or employee family member, contractor, agent, or business partner or a financial interest in the outcome of the trial

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 744 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of 2 doses of MVA-BN | 2 weeks after the second MVA-BN vaccination
  Titer of serum neutralizing antibodies against vaccinia virus as measured by plaque reduction neutralization tests (PRNTs)
Number of Participants with Serious Adverse Events (SAE) | From vaccination through study termination, up to 7 months
  Number and percentage of study participants reporting any serious adverse events at any time during the trial period
Number of Participants with Adverse Events of Special Interest (AESI) | From vaccination through study termination, up to 7 months
  Number and percentage of study participants reporting any Adverse Events of Special Interest (AESI)
Number of Participants with Medically Attended Adverse Events (MAAE) | From vaccination through study termination, up to 7 months
  Number and percentage of study participants reporting any Medically Attended Adverse Events (MAAE)
Number of Participants with a Grade 3 or higher adverse event (AE) | The day of or within 28 days after either vaccination
  Number and percentage of study participants reporting any grade 3 or higher unsolicited adverse event (AE) assessed as related to trial vaccine
Number of Participants with Solicited Local AE | The day of or within 7 days after either vaccination
  Number and percentage of study participants reporting any solicited local AE (pain, swelling, pruritus, erythema, induration)
Number of Participants with Solicited Systemic AE (body temperature, headache, fatigue, myalgia, nausea, chills) | The day of or within 7 days after either vaccination
  Number and percentage of study participants reporting any solicited systemic AE (body temperature, headache, fatigue, myalgia, nausea, chills)
Number of Participants with Unsolicited AE | The day of or within 28 days after either vaccination
  Number and percentage of study participants reporting any unsolicited AE

SECONDARY OUTCOMES:
Titer of Serum Neutralizing Antibodies against Vaccinia Virus | 4 weeks after the first MVA-BN vaccination and 6 months after the last MVA-BN vaccination
  GMTs of serum neutralizing antibodies against vaccinia virus as measured by PRNT
Seroconversion in Neutralizing Antibodies | 4 weeks after the first MVA-BN vaccination, 2 weeks and 6 months after the second MVA-BN vaccination
  Percentage of participants with seroconversion in neutralizing antibodies against vaccinia virus as determined by PRNT. Seroconversion is defined as either the appearance of antibody titer at or above the lower limit of quantitation [LLOQ] for participants with baseline values below the LLOQ or doubling or more of the antibody titer compared to baseline for participants with a baseline antibody titer at or above the LLOQ
Titer of Total Antibodies against Vaccinia Virus | 4 weeks after the first MVA-BN vaccination, 2 weeks and 6 months after the second MVA-BN vaccination
  GMTs of total antibodies against vaccinia virus as determined by enzyme-linked immunosorbent assay (ELISA)
Seroconversion in Total Antibodies against Vaccinia Virus | 4 weeks after the first MVA-BN vaccination, 2 weeks and 6 months after the second MVA-BN vaccination
  Percentage of participants with seroconversion in total antibodies against vaccinia virus as determined by ELISA Seroconversion is defined as either the appearance of total antibody at or above the LLOQ for participants with baseline values below the LLOQ, or a 4-fold increase of total antibodies against vaccinia virus compared to pre-immunization baseline values for participants with baseline values at or above the LLOQ

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Accellacare and McFarland Clinic, Ames, Iowa
  - Johnson County ClinTrials, LLC, Lenexa, Kansas
  - Rochester Clinical Research, Inc, Rochester, New York
  - Accellacare of Cary - Cary Medical Group, Cary, North Carolina
  - Accellacare Research of Salisbury, Salisbury, North Carolina
  - Accellacare of Charleston, Mt. Pleasant, South Carolina
  - Accellacare - Knoxville, Knoxville, Tennessee
  - Avacare, Austin, Texas
  - Avacare, Fort Worth, Texas
  - Velocity Clinical Research, Suffolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided